CLINICAL TRIAL: NCT00355394
Title: Treatment of Acute Migraine Headache in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2006-4-4755
Record Dates: First submitted 2006-07-19; First posted 2006-07-21 (Estimated); Results first posted 2013-08-30 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-10

CONDITIONS: Migrainous Headache
MeSH Terms: conditions — Migraine Disorders | interventions — Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Standard care including intravenous fluid, but no metoclopramide.
  Interventions: Other: Placebo
- Metoclopramide (Active Comparator): Standard care including intravenous fluid PLUS metoclopramide.
  Interventions: Drug: Metoclopramide

INTERVENTIONS:
Drug: Metoclopramide — Intravenous bolus administration.
  Other Names: Reglan
  Arms: Metoclopramide
Other: Placebo — Standard care including intravenous fluid, but no metoclopramide.
  Arms: Placebo

SUMMARY:
Migraine is common in children and is one of the most common etiologies of headache leading to emergency room presentation in children. Despite this, few studies have investigated the treatment of acute migraine headache in the emergency room. We will perform a prospective, double-blind, placebo-controlled study of metoclopramide versus placebo in the treatment of acute migraine headache. The primary outcome will be the number of subjects headache free at two hours.

DETAILED DESCRIPTION:
Migraine is common in children and is one of the most common etiologies of headache leading to emergency room presentation of children [1-3]. Despite the high prevalence, there have been few pediatric studies of the acute treatment of migraine headache. Anti-dopaminergic medications such as metoclopramide are often considered first line medications in the emergency room treatment of acute migraine [personal communication with Children's Hospital of Philadelphia Emergency Department physicians], but only two pediatric studies guide this clinical management. One was a retrospective, uncontrolled, descriptive study [4] and one was a prospective, double-blind study that compared an anti-dopaminergic medication to a different medication but did not include a control group [5]. More rigorous studies are needed to determine whether commonly utilized anti-dopaminergic medications are efficacious.

We will perform a prospective, randomized, double-blind placebo controlled study of the acute treatment of pediatric migrainous headache with metoclopramide.

Primary Objective The primary objective of the study is to determine whether metoclopramide added to standard care [intravenous (iv) hydration, darkened room] is superior to placebo and standard care in resolving acute migraine headache intensity within two hours in children aged 8 to 18 years presenting to the emergency department (ED).

Secondary Objectives:

1. Determine whether metoclopramide added to standard care (iv hydration, darkened room) is superior to placebo and standard care in resolving acute migraine headache intensity within one hour in children aged 8 to 18 years presenting to the emergency department.
2. Determine whether metoclopramide added to standard care (iv hydration, darkened room) is superior to placebo and standard care in resolving acute migraine headache intensity at 24 hours in children aged 8 to 18 years presenting to the emergency department.

Study Design:

The study is a prospective, randomized, double-blind, placebo-controlled study of metoclopramide versus placebo. Subjects may receive up to two doses of study medication one hour apart.

Children who present to the emergency department with migraine headache based on International Classification of Headache Disorders (ICHD) criteria will be eligible for enrollment. A standard assessment form will be sued to ensure children meet ICHD criteria. Children will then be randomized to receive either metoclopramide or placebo (intravenous fluid injection). Both patients and the study investigator performing assessments will be blind as to group assignment, while the Emergency Department physician will be aware of group assignment (acting as the pharmacist) so that if problems arise they can be evaluated and treated as clinically indicated. Assessment of headache and associated features will occur at one hour. If the child is not headache free, they will receive a second dose of either metoclopramide or placebo. If they received metoclopramide initially the second dose will be metoclopramide, and if they received placebo initially the second dose will be placebo. Assessment of headache and associated features will occur again at two hours. This marks the primary endpoint, as our primary objective is to determine whether metoclopramide is superior to placebo in making patients headache free at two hours.

Headache recurrence will be assessed at 24 hours.

Subject Population:

Children will be recruited from the Emergency Department. Consent and assent will be obtained as described in the protocol.

Number of Subjects:

All subjects will be recruited from the Emergency Department of a single institution. Sample size calculation suggests we will need 44 subjects for analysis.

Study Duration The total duration of the study is one day for each subject. The maximum time spent in the Emergency Department will be six hours. We expect subject enrollment to take approximately six months.

Study Phases:

1. Screening Phase: Upon presentation to the Emergency Department, patients diagnosed with migrainous headache based on International Classification of Headache Disorders criteria will be considered for enrollment. If they meet inclusion and exclusion criteria they will be consented/assented and enrolled in the study.
2. Basic Information Collection Basic demographic information, medical history, psychological/psychiatric history past headache history, and information regarding the current headache will be gathered.
3. Double-Blind Study Subjects will be randomized to receive metoclopramide or placebo in a double blind study. Baseline headache and associated symptom data will be gathered. Assessments will be performed at one hour and two hours. The two hour assessment is the primary endpoint. If the headache has not resolved, the cross-over will occur. Children who received metoclopramide initially will receive a placebo injection and, if needed, a second injection one hour later. Children who received placebo initially will receive metoclopramide and, if needed, a second injection one hour later. Headache assessments will be performed one and two hours after the cross-over.
4. Follow-up Phase Patients will rate their headache intensity and associated symptoms at one day in order to assess for recurrence.

Efficacy Evaluations:

Efficacy will be judged hourly after each medication (or placebo administration). Efficacy in reducing headache intensity will be judged on a 0-10 point numerical rating scale. The primary measure of efficacy will be headache freedom (rating of zero). Secondary measures will be improvement in headache intensity that is clinically relevant (6 point improvement) or improvement that is measurable (3 point improvement), improvement in associated symptoms (based on a 4 point categorical scale), or improvement in disability (based on a 4 point categorical scale).

Safety Evaluations:

All subjects entered in the study will be included in safety analysis. The frequency and descriptions of all adverse events will be summarized. Any serious adverse events will be described in detail.

Statistical And Analytic Plan:

Based on prior studies, we estimate a metoclopramide efficacy of 80% and placebo rate of 35%. Sample size and power calculations using an alpha value of 0.05 and power of 0.8 demonstrate that we will need to enroll 44 patients in the study. Subjects who drop out due to need for faster rescue medication will be maintained in the analysis which will be performed in an intent-to-treat manner.

ELIGIBILITY:
Inclusion Criteria:

1. Males or Females age 8-18 years
2. Girls 11 years or older must have a negative urine/serum pregnancy test.
3. Diagnosis of pediatric migrainous headache. The criteria for pediatric migraine headache based on the most recent ICHD criteria are listed below. The requirement of 5 attacks (A) will not be required for this study, this making the diagnosis migrainous headache. As described elsewhere in the protocol, this change is required to make the study applicable to ED patients who require treatment before five attacks have occurred.

Exclusion Criteria:

1. Evidence that headache is due to a secondary underlying disorder based on history or physical examination.
2. Pregnant or lactating females.
3. Any investigational drug use within 30 days.
4. Known to have a contraindication to metoclopramide or valproic acid such as pregnancy, liver disease, hematologic disease, or metabolic disease.
5. Have used metoclopramide (or other antidopaminergic medications) or valproic acid within two days of presentation.
6. Severe developmental disorders or mental retardation if insufficient information can be obtained to make a clear diagnosis of migraine or judge headache severity.
7. If patients re-present to the ED, they can not be re-enrolled.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2006-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas S Abend, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited from tertiary care emergency department (ED). N=31.
Groups:
- Placebo: Placebo group received standard care including IVF but not metoclopramide.
- Metoclopramide: Metoclopramide group received standard care including IVF and also IV metoclopramide.
Period: Overall Study
Arm/Group | Placebo | Metoclopramide
Started | 15 | 16
Completed | 15 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Metoclopramide: Metoclopramide group received standard care including IVF AND metoclopramide.
- Total: Total of all reporting groups
Arm/Group | Placebo | Metoclopramide | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 16 | 31
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.8 (3.1) | 12.9 (2.4) | 11.9 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 6 | 8 | 14
Region of Enrollment [Number; unit: participants]
  United States | 15 | 16 | 31

OUTCOME MEASURES:

1. Primary Outcome: The Number of Subjects With a Numeric Rating Scale Score (NRS) of Zero at Two Hours.
Description: The NRS is a 0 to 10 point scale with 0 representing no headache and 10 representing severe headache.
Time Frame: 2 hours
Population: All participants included.
Measure: Number; unit: participants
Groups:
- Placebo: Placebo
- Metoclopramide: Metoclopramide
Arm/Group | Placebo | Metoclopramide
Number analyzed (Participants) | 15 | 16
participants | 5 | 12
Statistical Analysis 1: Comparison: Placebo vs Metoclopramide; Test type: Superiority or Other; p = 0.03, Fisher Exact

2. Secondary Outcome: The Number of Subjects With a NRS Score of Zero at One Hour.
Description: The NRS is a 0 to 10 point scale with 0 representing no headache and 10 representing severe headache.
Time Frame: 1 hour
Population: All participants included.
Measure: Number; unit: participants
Arm/Group | Placebo | Metoclopramide
Number analyzed (Participants) | 15 | 16
participants | 1 | 9
Statistical Analysis 1: Comparison: Placebo vs Metoclopramide; Test type: Superiority or Other; p = 0.02, Fisher Exact

3. Secondary Outcome: The Number of Subjects With a NRS Score of Zero at 24 Hours.
Description: The NRS is a 0 to 10 point scale with 0 representing no headache and 10 representing severe headache.
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | Placebo | Metoclopramide
Number analyzed (Participants) | 15 | 16
participants | 4 | 7
Statistical Analysis 1: Comparison: Placebo vs Metoclopramide; Test type: Superiority or Other; p = 0.46, Fisher Exact

4. Secondary Outcome: Change in Headache Intensity as Measured by the NRS Score From Baseline to the One Hour Assessment.
Description: The NRS is a 0 to 10 point scale with 0 representing no headache and 10 representing severe headache.
Time Frame: 1 hours
Population: All participants included.
Measure: Mean (Standard Deviation); unit: NRS Score
Arm/Group | Placebo | Metoclopramide
Number analyzed (Participants) | 15 | 16
NRS Score | -2.5 (2.5) | -6.8 (3.1)
Statistical Analysis 1: Comparison: Placebo vs Metoclopramide; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change in Headache Intensity as Measured by the NRS Score From Baseline to the Two Hour Assessment.
Description: The NRS is a 0 to 10 point scale with 0 representing no headache and 10 representing severe headache.
Time Frame: 2 hours
Measure: Median (Standard Deviation); unit: NRS Score
Arm/Group | Placebo | Metoclopramide
Number analyzed (Participants) | 15 | 16
NRS Score | -4.9 (2.8) | -7.8 (2.1)
Statistical Analysis 1: Comparison: Placebo vs Metoclopramide; Test type: Superiority or Other; p = 0.01, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Change in Headache Intensity as Measured by the NRS Score From Baseline to the 24 Hour Assessment.
Description: The NRS is a 0 to 10 point scale with 0 representing no headache and 10 representing severe headache.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: NRS Score
Arm/Group | Placebo | Metoclopramide
Number analyzed (Participants) | 15 | 16
NRS Score | -4.5 (2.9) | -5.6 (3.3)
Statistical Analysis 1: Comparison: Placebo vs Metoclopramide; Test type: Superiority or Other; p = 0.50, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Placebo | Metoclopramide
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 0/15 | 0/16

LIMITATIONS AND CAVEATS:
Study was performed in tertiary care setting and may not be generalizable to all settings. Small number of subjects (n=31). None admitted or received additional rescue medication, suggesting most severely affected may not have been enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No